CLINICAL TRIAL: NCT00969618
Title: Long-Term, Open-Label Safety and Efficacy Study of Atomoxetine Hydrochloride in Adult Patients With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: A Long Term Follow-Up Study for Asian Adult Patients With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12397; B4Z-JE-LYEK (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Results first posted 2012-12-12 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-11

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atomoxetine (Experimental)
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine — 40-120 milligrams/day (mg/day) taken by mouth, once a day for 48 weeks
  Other Names: LY139603; Strattera

SUMMARY:
The purpose of this study is to assess long-term safety and tolerability in adult patients who have completed a previous atomoxetine study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed the B4Z-JE-LYEE study (NCT00962104) and signed the Informed Consent Document (ICD).
* Patients must have been judged by the investigator to be reliable to keep appointments for clinic visits and all tests, including venipuncture and examinations, required by the protocol.
* Patients must possess an educational level and degree of understanding of the language of their country that enables them to communicate suitably with the investigator and study coordinator.

Exclusion Criteria:

* Patients who meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision criteria for current anxiety disorder and also patients who require anti-anxiety drug therapy within previous study except for those taking benzodiazepines analogs for anxiety. The dosage of diazepam equivalents should not be more than 5 milligrams/day (mg/day).
* Patients who, in the opinion of the investigator, are at serious suicidal risk or serious risk of harming others, or whose score for Item 11 on the Hamilton Depression Rating Scale-17 items is equal or more than 2 at randomization or screening.
* Patients with significant medical conditions that are likely to become unstable during the trial or would likely be destabilized by treatment with atomoxetine or require treatment with excluded medications.
* Patients with a history of allergy to atomoxetine, severe allergies to more than 1 class of medications, or multiple adverse drug reactions.
* Patients who have received treatment within the past 30 days with a drug that has not received regulatory approval for any indication at the time the informed consent document is obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2009-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- Japan (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukushima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atomoxetine
Started | 211
Completed | 133
Not Completed | 78
Not completed — Adverse Event | 29
Not completed — Entry Criteria Not Met | 3
Not completed — Lack of Efficacy | 2
Not completed — Lost to Follow-up | 7
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 9
Not completed — Withdrawal by Subject | 27

BASELINE CHARACTERISTICS:
Arm/Group | Atomoxetine
Number analyzed (Participants) | 211
Age Continuous [Mean (Standard Deviation); unit: years] | 32.6 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105
  Male | 106
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 211
Region of Enrollment [Number; unit: participants]
  Japan | 211

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Leading to Discontinuation
Time Frame: Baseline through 48 weeks
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: participant
Arm/Group | Atomoxetine
Number analyzed (Participants) | 211
participant | 29 [9.1 to 18.4]

2. Secondary Outcome: Mean Change From Baseline to 48 Weeks Endpoint in the Conners' Adult Attention-Deficit Hyperactivity Disorder Rating Scale-Investigator Rated: Screening Version-Japanese (CAARS-Inv:SV-J)
Description: CAARS-Inv:SV-J is a 30-item scale containing 3 subscales: inattention (9 items), hyperactivity/impulsivity (9 items), and attention deficit hyperactivity disorder (ADHD) Index (12 items). Each item is scored 0-3 (0=not at all/never; 1=just a little/once in a while; 2=pretty much/often; 3=very much/very frequently). Total ADHD symptoms score=sum of the inattention subscales (scores range from 0-27) and hyperactivity/impulsivity subscales (scores range from 0-27) with a total score range of 0-54. The ADHD Index scores range from 0-36. Higher scores indicate greater impairment.
Time Frame: Baseline, 48 weeks
Population: All participants who received at least one dose of study drug, and had a baseline and at least one post-baseline CAARS measurement. Last observation carried forward (LOCF) principle was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 211
units on a scale
  Total ADHD Symptoms Score | -7.3 (8.1)
  Inattention Subscale Score | -4.6 (5.1)
  Hyperactivity/Impulsivity Subscale Score | -2.7 (4.2)
  ADHD Index Subscale Score | -5.0 (5.9)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-value is for total ADHD symptoms score
Statistical Analysis 2: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-value is for inattention subscale score
Statistical Analysis 3: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-value is for hyperactivity/impulsivity subscale score
Statistical Analysis 4: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-value is for ADHD index subscale score

3. Secondary Outcome: Mean Change From Baseline to 48 Weeks Endpoint in the Adult Attention-Deficit/Hyperactivity Disorder Quality of Life (AAQoL)-29 Scores
Description: AAQoL is a 29 items participant completed questionnaire rated on a 5-point Likert scale from 1 (Not at all/ Never) to 5 (Extremely/Very Often). AAQoL total (all 29 items) and 4 subscale scores: Life Productivity (11 items); Psychological Health (6 items); Life Outlook (7 items); Relationships (5 items). Total score is computed by (1) reversing scores for all items except the 7 items in the Life Outlook subscale; (2) transforming scores to 0-100 scale (1=0; 2=25; 3=50; 4=75; 5=100); (3) summing item scores and dividing by the item count. Higher total scores indicate better quality of life.
Time Frame: Baseline, 48 weeks
Population: All participants who received at least one dose of study drug, and had a baseline and at least one post-baseline AAQoL measurement. Last observation carried forward (LOCF) principle was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 206
units on a scale | 4.46 (13.44)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test

4. Secondary Outcome: Mean Change From Baseline to 48 Weeks Endpoint in the Behavior Rating Inventory of Executive Function -Adult (BRIEF-A) Version: Self Report (BRIEF-A:Self Report )
Description: A 75-item standardized self-reported measure comprised of 3 subscales. Each item is rated on a 3-point Likert scale: 1 (behavior never observed) to 3 (behavior often observed). Global executive composite (GEC) subscale rates participant's GEC in everyday environment (75- 225 total score). Behavioral regulation subscale measures participant's control over behavior (30-90 total score). Metacognition subscale assesses systematic problem-solving ability while sustaining these task-completion efforts in active working memory (40-120 total score). Higher subscale ratings indicate greater perceived impairment.
Time Frame: Baseline, 48 weeks
Population: All participants who received at least one dose of study drug, and had a baseline and at least one post-baseline BRIEF-A self report measurement. Last observation carried forward (LOCF) principle was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 206
units on a scale
  GEC Subscale Score | -10.4 (21.3)
  Behavioral Regulation Subscale Score | -3.6 (9.2)
  Metacognition Subscale Score | -6.8 (13.6)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-value is GEC subscale score
Statistical Analysis 2: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-value is for behavioral regulation subscale score
Statistical Analysis 3: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-value is for metacognition subscale score

5. Secondary Outcome: Mean Change From Baseline to 48 Weeks Endpoint in Comorbid, Anxiety Symptoms, as Measured by Hamilton Anxiety Rating Scale-14 (HAMA-14) Items
Description: The HAMA-14 instrument consists of 14 items that provide an overall measure of general anxiety, including psychic anxiety and somatic anxiety. This instrument is completed by the clinician based on his or her assessment of the participant. Each item is rated on a 5-point scale of 0 (absent) to 4 (very severe). Total score is the sum of the 14 items and ranges from 0 (normal) to 56 (severe). Higher scores indicate greater anxiety.
Time Frame: Baseline, 48 weeks
Population: All participants who received at least one dose of study drug, and had a baseline and at least one post-baseline HAMA-14 measurement. Last observation carried forward (LOCF) principle was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 198
units on a scale | 0.3 (3.1)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.200, Paired t-test

6. Secondary Outcome: Mean Change From Baseline to 48 Weeks Endpoint in Clinical Global Impressions-Attention-Deficit/Hyperactivity Disorder-Severity (CGI-ADHD-S)
Description: The CGI-ADHD-S is a single-item rating of the clinician's assessment of the overall severity of the participant's ADHD symptoms in relation to the clinician's total experience with ADHD participants. CGI-ADHD-S measures severity of the participant's overall severity of ADHD symptoms: 1 (normal, not at all ill) to 7 (among the most extremely ill participants).
Time Frame: Baseline, 48 weeks
Population: All participants who received at least one dose of study drug, and had a baseline and at least one post-baseline CGI-ADHD-S measurement. Last observation carried forward (LOCF) principle was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 211
units on a scale | -0.8 (1.0)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test

7. Secondary Outcome: Mean Change From Baseline to 48 Weeks Endpoint in the Behavior Rating Inventory of Executive Function-Adult (BRIEF-A) Version: Informant Scores (BRIEF-A:Informant Scores)
Description: Third-party observer of participant completes 75-item scale. Comprised of 3 subscales. Each item rated on 3-point Likert scale: 1 (behavior never observed) to 3 (behavior often observed). Global executive composite (GEC) subscale rates participant's GEC in everyday environment (75-225 total score). Behavioral regulation subscale measures participant's control over behavior (30-90 total score). Metacognition subscale assesses systematic problem-solving ability while sustaining these task-completion efforts in active working memory (40-120 total score). Higher subscale ratings indicate greater perceived impairment.
Time Frame: Baseline, 48 weeks
Population: All participants who received at least one dose of study drug, and had a baseline and at least one post-baseline BRIEF-A Informant scores measurement. Last observation carried forward (LOCF) principle was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 148
units on a scale
  GEC Subscale Score (n=146) | -8.5 (22.5)
  Behavioral Regulation Subscale Score (n=148) | -2.9 (10.0)
  Metacognition Subscale Score (n=147) | -5.5 (14.0)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-value is for GEC subscale score
Statistical Analysis 2: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-value is for behavioral regulation subscale score
Statistical Analysis 3: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-value is for metacognition subscale score

8. Secondary Outcome: Mean Change From Baseline to 48 Weeks Endpoint in Comorbid, Depressive Symptoms, as Measured by Hamilton Depression Rating Scale-17 (HAMD-17) Items
Description: The HAMD-17 instrument consists of 17 items used to assess the severity of depression and its improvement during the course of therapy. This instrument is completed by the clinician based on his or her assessment of the participant. Each item was evaluated and scored using either a 5-point scale of 0 (not present) to 4 (very severe) or a 3-point scale of 0 (not present) to 2 (marked). The total score is the sum of the scores from HAMD-17 Items 1 through 17 and ranges from 0 (not at all depressed) to 52 (severely depressed). Higher scores indicate greater symptom severity.
Time Frame: Baseline, 48 weeks
Population: All participants who received at least one dose of study drug, and had a baseline and at least one post-baseline HAMD-17 measurement. Last observation carried forward (LOCF) principle was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 198
units on a scale | 0.2 (2.9)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.384, Paired t-test

ADVERSE EVENTS:
Arm/Group | Atomoxetine
Serious Adverse Events (participants affected / at risk) | 5/211
Other Adverse Events (participants affected / at risk) | 180/211
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=211)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Infectious peritonitis (Infections and infestations) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=211)
Palpitations (Cardiac disorders) | 14 (14)
Tachycardia (Cardiac disorders) | 11 (11)
Abdominal discomfort (Gastrointestinal disorders) | 11 (15)
Constipation (Gastrointestinal disorders) | 16 (18)
Nausea (Gastrointestinal disorders) | 90 (121)
Vomiting (Gastrointestinal disorders) | 13 (29)
Thirst (General disorders) | 28 (33)
Seasonal allergy (Immune system disorders) | 11 (11)
Nasopharyngitis (Infections and infestations) | 67 (100)
Decreased appetite (Metabolism and nutrition disorders) | 20 (21)
Headache (Nervous system disorders) | 31 (48)
Somnolence (Nervous system disorders) | 19 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days